CLINICAL TRIAL: NCT03751826
Title: Peer Delivery of HIV Self-Screening to Support Linkage to HIV Prevention in Rural KwaZulu-Natal, South Africa: A Cluster Randomized Control Trial
Brief Title: Peer Delivery of HIV Self Test to Improve Linkage to HIV Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Collaborators: Africa Health Research Institute (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15990
Record Dates: First submitted 2018-11-07; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: HIV
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The unit of randomisation will be pairs of peer navigators: 21 pairs of peer navigators will be randomised to 3 arms: two intervention arms, and standard of care (7 pairs per arm).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Incentivised network delivery HIV-ST (Experimental): Peer-navigators will use respondent-driven sampling to distribute HIV-ST kits through 'seeds'. Each 'seed' (female aged 18-24 years) will receive a session on HIV prevention, the importance of sexual health, the benefits of HIV testing PrEP and ART, and a demonstration of HIV self-screening. Seeds will be asked to recruit females aged 18-24 years and given 5 uniquely numbered incentivized recruitment coupons with HIV-ST kits to pass on to their peers. Individual who return the coupons will undergo the same procedure as the seeds above and the individual who handed out the coupon will receive a sum of $1.5 in airtime per friend who returns the coupon. The packs include referral slips with information on how to link to HIV community-based confirmatory testing, HIV treatment and PrEP.
  Interventions: Other: Incentivised network delivery of HIV-ST
- Peer Navigator distributed HIV-ST (Experimental): Peer navigators will directly distribute HIV-ST kits to females aged 18-24 years over a period of six months. Each person recruited will receive a session from the peer-navigator on the HIV prevention services available, the importance of sexual health, the benefits of HIV testing PrEP and ART, and a demonstration of HIV-ST. The packs include referral slips with information on how to link to community-based HIV confirmatory testing, HIV treatment and PrEP.
  Interventions: Other: Peer navigator delivery of HIV-ST
- Standard of care (Active Comparator): Peer navigators will encourage females aged 18-24 years to test for HIV at clinics, and link to services/care. Each female aged 18-24 approached by a peer navigator will receive a session from the peer-navigator on the HIV prevention services available, the importance of sexual health, the benefits of HIV testing PrEP and ART, and a demonstration of HIV self-screening. They will then be given a referral slip for HIV testing through the clinic. The referral slips include information on how to link to community-based HIV confirmatory testing, HIV treatment and PrEP.
  Interventions: Other: standard of care

INTERVENTIONS:
Other: Incentivised network delivery of HIV-ST — Peer navigators are area based young community care givers, who support young people in their area in the uptake of multi-level HIV prevention provided through the department of health, social welfare and basic education, e.g. parenting support, gender-based violence interventions, safe spaces, mentoring, life-skills, and support around knowing and getting social entitlements and financial literacy. The peer navigators in the first intervention arm will encourage females aged 18-24 to use the HIV-ST to test for HIV themselves and in their peers and friends. They will be counselled to receive sexual and reproductive health services, contraception and condoms, HIV confirmatory testing and linkage to HIV care and prevention, including HIV Pre-Exposure Prophylaxis (PrEP), through referral slips to the study mobile clinical services.
  Arms: Incentivised network delivery HIV-ST
Other: Peer navigator delivery of HIV-ST — Peer navigators are area based young community care givers, who support young people in their area in the uptake of multi-level HIV prevention provided through the department of health, social welfare and basic education, e.g. parenting support, gender-based violence interventions, safe spaces, mentoring, life-skills, and support around knowing and getting social entitlements and financial literacy. The peer navigators in the second intervention arm will encourage females aged 18-24 to use the HIV-ST to test for HIV and then receive sexual and reproductive health services, contraception and condoms, HIV confirmatory testing and linkage to HIV care and prevention, including HIV Pre-Exposure Prophylaxis (PrEP), through referral slips to the study mobile clinical services.
  Arms: Peer Navigator distributed HIV-ST
Other: standard of care — Peer navigators are area based young community care givers, who support young people in their area in the uptake of multi-level HIV prevention provided through the department of health, social welfare and basic education, e.g. parenting support, gender-based violence interventions, safe spaces, mentoring, life-skills, and support around knowing and getting social entitlements and financial literacy. The peer navigators in the standard of care arm encourage females aged 18-24 to test for HIV, receive sexual and reproductive health services, contraception and condoms, and link to HIV care and prevention, including HIV Pre-Exposure Prophylaxis (PrEP), through referral slips to the study mobile clinical services.
  Arms: Standard of care

SUMMARY:
Hypothesis: HIV-Self-Test (HIV-ST) will allow peers or peer-networks to effectively and efficiently link older adolescent girls and young women into HIV prevention and care services.

Design: A cluster randomized control trial comparing two models of peer delivery of HIV-ST, through incentivized respondent driven peer networks and direct distribution by peer navigators compared to standard of care (referral to HIV testing, prevention and care services by peer navigators) in improving the uptake of HIV prevention and care amongst young women (18-24) living in the rural uMkhanyakude district of KwaZulu-Natal, South Africa.

Objectives:

1. To increase the knowledge of HIV status among young women aged 18-24 years old through distribution of HIV-ST through incentivized peer networks or direct distribution by peer navigators compared to peer navigators referring into HIV testing services.
2. To determine an increase in the rate of linkage among young women aged 18-24 to HIV prevention and treatment services facilitated by distribution of HIV-ST through incentivized peer networks or direct distribution by peer navigators compared to peer navigators referring into services.
3. To conduct a process evaluation of the acceptability, feasibility, and reach (out of school, recently migrant and living in remote areas) in linking 18-24-year-old women to HIV prevention and treatment services of HIV-ST distribution through incentivized peer networks, or direct distribution by peer navigators or peer navigators referring into services.
4. To measure the cost per 18-24-year-old linked to prevention and care through peer-led incentivized HIV-ST delivery system or direct distribution of HIV-SS by peer navigators, compared to peer navigator referring into services.

Primary Outcomes:

The difference between the rate of linkage within three months of 18-24 years old women to HIV confirmatory testing and pre-exposure prophylaxis (PrEP) eligibility screening if HIV-negative and antiretroviral treatment (ART) starting if HIV-positive. It will be between the two peer-delivery approaches to HIV-ST distribution (incentivized HIV-ST delivery through peer network and direct distribution of HIV-ST by peer navigators) compared to standard of care (peer navigator referral to HIV testing, treatment and prevention services). Rate is defined as the number of linkages per month of peer navigator outreach activity.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Aged 18-24 years
* Not currently on ART
* Provide written informed consent

Exclusion Criteria:

* Under 18 years or older than 24 years
* Participants not willing to consent or unable to provide informed consent
* Males
* Currently on ART

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — everyone is eligible to receive the HIV self screen, but the primary outcome of linkage to care is only measured in self identified females aged aged 18-24 years
Enrollment: 2000 (Estimated)
Dates: Start 2019-01-14 (Estimated); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of linkage among women ages 18-24 years to HIV prevention services. | within 3 months of receiving the intervention
  The rate of linkage per month of peer navigator activity to a confirmatory testing and pre-exposure prophylaxis (PrEP) eligibility screening if HIV-negative and antiretroviral treatment (ART) starting if HIV-positive.

SECONDARY OUTCOMES:
The number of linkages per 100 clinic referral slips distributed per arm; | within 3 months of receiving the intervention.
  The number of linkages to a confirmatory testing and pre-exposure prophylaxis (PrEP) eligibility screening if HIV-negative and antiretroviral treatment (ART) starting if HIV-positive per 100 clinic referral slips distributed per arm.
The change in proportion of all residents (men and women) aged 18-24 years who are aware of HIV-SS and who have used HIV-SS over time | 12 months following intervention end date
  Using routine annually collected data from the surveillance area
Comparison of the difference per study area in the proportion of 18-24 year olds who report knowledge of HIV status and uptake of ART, PrEP and voluntary medical male circumcision (VMMC) | 12 months following intervention end date
  Using routine annually collected data from the surveillance area
Comparison of the pattern of recruitment per arm of study | 12 months following intervention end date
  The proportion of hard to reach adolescent girls and young women (aged 18-24 years) - defined as out of school, recently migrated and those who live in remote areas - linked to care in the three arms of study
Comparison of costs per case linked to PrEP eligibility assessment (HIV-) and cost per case started on ART (HIV+) in intervention and control arms | 6 months study implementation period
  To establish costs, we will use both a bottom-up ingredient-based costing approach and a top-down costing approach using the study budgets and expenditure reports.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Shahmanesh, MRCP PhD, Principal Investigator — University College London and Africa Health Research Institute

IPD SHARING:
Plan to Share IPD: Yes
We are committed to open access data and so we have developed systems to support safe sharing. The data will be managed within the AHRI Data Management Centre, where they are linked to population data. The data is supplied to investigators de-identified.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The study team will have exclusive use of the data for 2 years after the study and/or once the primary analysis of the study has been published, whichever comes first. Data may be made available sooner at the discretion of the investigators, where this does not conflict with the publication plans for the study. After the period of exclusive use, data will be made available to potential new users on request.
Access Criteria: The data custodian has the administrative control over granting access to the data to researchers. Anonymized electronic quantitative datasets will be archived and made available to interested external researchers. Requests for data sharing are reviewed by the data custodian and a Data Sharing committee at AHRI. All AHRI staff are bound by the AHRI Data Access Policy, which prohibits any sharing of data with third parties, unless a formal Data Use Agreement has been signed with the third party. The Data Use Agreement defines the analyses to be undertaken. If approved the study would have to undergo relevant IRB and ethical review processes.

REFERENCES:
- [Derived] Shahmanesh M, Mthiyane TN, Herbsst C, Neuman M, Adeagbo O, Mee P, Chimbindi N, Smit T, Okesola N, Harling G, McGrath N, Sherr L, Seeley J, Subedar H, Johnson C, Hatzold K, Terris-Prestholt F, Cowan FM, Corbett EL. Effect of peer-distributed HIV self-test kits on demand for biomedical HIV prevention in rural KwaZulu-Natal, South Africa: a three-armed cluster-randomised trial comparing social networks versus direct delivery. BMJ Glob Health. 2021 Jul;6(Suppl 4):e004574. doi: 10.1136/bmjgh-2020-004574. PMID 34315730
- [Derived] Adeagbo OA, Mthiyane N, Herbst C, Mee P, Neuman M, Dreyer J, Chimbindi N, Smit T, Okesola N, Johnson C, Hatzold K, Seeley J, Cowan F, Corbett L, Shahmanesh M. Cluster randomised controlled trial to determine the effect of peer delivery HIV self-testing to support linkage to HIV prevention among young women in rural KwaZulu-Natal, South Africa: a study protocol. BMJ Open. 2019 Dec 23;9(12):e033435. doi: 10.1136/bmjopen-2019-033435. PMID 31874891